CLINICAL TRIAL: NCT01832701
Title: Coffee and Oxidative Stress During Exercise in Healthy Humans
Brief Title: Coffee, Exercise, and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 10.38.MET
Record Dates: First submitted 2013-04-08; First posted 2013-04-16 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
MeSH Terms: interventions — Coffee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- coffee (Experimental): 4 cups of soluble coffee per day (2.5g per cup)
  Interventions: Other: Placebo comparator
- Maltodextrine with caffeine (Placebo Comparator): 4 cups per day containing 2.5 g of product each
  Interventions: Other: Coffee

INTERVENTIONS:
Other: Coffee — coffee versus placebo
  Arms: Maltodextrine with caffeine
Other: Placebo comparator — maltodextrine with caffeine
  Arms: coffee

SUMMARY:
Coffee is one of the most widely consumed beverages. It contains polyphenols (chlorogenic acids) and bioavailability of these bioactive compounds is now somewhat well understood. In addition, chlorogenic acids are known to be antioxidants in the cup, but reliable evidence remains to be observed in vivo. The objective of this trial is to understand if regular (14d) coffee intake may be beneficial on biomarkers of oxidative damage measured in urine and plasma after an acute stress caused by exercise.

DETAILED DESCRIPTION:
Coffee is one of the most widely consumed beverages. It contains polyphenols (chlorogenic acids) and bioavailability of these bioactive compounds is now somewhat well understood. However, even if chlorogenic acids are known to be antioxidants in the cup, reliable evidence remains to be observed in vivo.

After medical examination and approval, subjects will undergo 2 periods of 21 days. The first 7 days will consist of a dietary restriction to lower the polyphenols intake. Then subjects will drink at random one of the three treatments for 14 days (4 cups/day). Blood and urine samples will be collected throughout the study to evaluate in vivo effects on oxidative biomarkers. Furthermore, at day 21, subjects will undergo a physical regimen to increase acutely and transiently their oxidative damage. Blood and urine samples collected throughout this challenge will allow us to evaluate the effect of coffee intake in reducing oxidative damage created by exercise compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal and overweight subjects (BMI 19 - 29), with lean mass below the 90th percentile value
* Coffee drinkers with an average consumption of 1-3 cups per day
* Having given informed consent
* VO2 max as a function of age and gender, not higher than the values below:

Max oxygen uptake (VO2max, in ml/kg/min) in non athletes Age Males Females 20-29 49 41 30-39 47 39 40-49 45 37

Exclusion Criteria:

* Digestive (intestinal, gastric, hepatic or pancreatic), renal or metabolic disease, as determined by the medical (screening) visit and a blood chemistry analysis (glucose, cholesterol, LDL, HDL, triglycerides, aspartate transaminase (ASAT), Alanine transaminase (ALAT), C reactive Protein (CRP), creatinin)
* Subjects at cardio-vascular risk rated as intermediate or high (according to the Swiss Society of Cardiology, lipids group (www.agla.ch/p11-1-2.html), meaning those who show at least one of the following criteria:

  * History of coronary disease / atherosclerosis
  * Diabetes
  * High level of risk (familial hypercholesterolemia, hyperlipoproteinemia type III, hypertension)
  * Metabolic syndrome defined by the presence of at least 3 out of the following criteria :

Abdominal circumference > 102 cm in men, > 88 cm in women Fasting triglycerides ≥ 1.7 mmol/l HDL-cholesterol < 1.0 mmol/l in men, < 1.3 mmol/l in women Systolic arterial blood pressure ≥ 130 mm Hg and/or diastolic arterial blood pressure ≥ 85 mm Hg Plasma glucose ≥ 6.1 mmol/l

* Anemia (Erythrocytes < 4.6 T/l (male) or < 4.2 T/l (women); Hemoglobin Hb < 13 g/dl (male) or Hb < 12 g/dl (women); Hematocrit Ht < 40% (male) or Ht < 37% (women); sera iron < 0.6 mg/l or plasma ferritin < 120 microg /l (male) or < 60 microg/l (non menopausal women)
* Troubles of hemostasis as determined by platelets number, prothrombin time and activated partial thromboplastin time
* Have had a gastrointestinal surgery, except appendicectomy
* Pregnancy
* History of food or medication allergy
* Have a regular consumption of medication (only those impacting oxidative stress biomarkers (eg. impacting the metabolism of lipids / LDL / VLDL), oral contraception excepted)
* Have taken antibiotic therapy within the last 3 months
* Smokers (more than 5 cigarettes per day)
* Having given blood within the last month, or willing to make a blood donation until one month following the end of the study
* Have a high alcohol consumption (more than 2 drinks/day)
* Taking more than 3 cups of coffee per day
* Consumption of illicit drugs
* Subject who cannot be expected to comply with the study procedures, including consuming the test products.
* Currently participating or having participated in another clinical trial during the last month prior to the beginning of this study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
oxidative stress | Change in oxidative stress from baseline to the last day of a 14-day period of product intake
  Oxidative stress will be assessed though urine beta-isoprostane measurements

SECONDARY OUTCOMES:
Bioavailability of coffee antioxidative compounds | Change in urine phenolic and chlorogenic acids from baseline to the last day of a 14-day period of product intake
  Measures of phenolic and chlorogenic acids in urine

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Beaumont, MD, Principal Investigator — Clinical Development Unit / Metabolic Unit
Locations (1):
- Clinical Development Unit / Metabolic Unit, Lausanne, Switzerland